CLINICAL TRIAL: NCT03167866
Title: The Influence of Motivational Text Messages on Glycemic Control and Healthy Lifestyle Choices in Patients With Diabetes
Brief Title: Effect of Motivation Text Messages on Diabetes Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 66666
Record Dates: First submitted 2017-04-26; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization will be by study personell that is not in contact with participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): DM patients who receive a weekly informational Short Message Service (SMS) by phone for 26 weeks. informational SMS
  Interventions: Behavioral: informational SMS
- test group (Experimental): DM patients who receive a weekly motivational Short Message Service (SMS) for 26 weeks. motivational SMS
  Interventions: Behavioral: motivational SMS

INTERVENTIONS:
Behavioral: motivational SMS — the participant receives a weekly text message that is aimed to increase motivation
  Arms: test group
Behavioral: informational SMS — the participant a weekly text message that is provides information on improving lifestyle
  Arms: control group

SUMMARY:
The investigators will examine the influence of increasing motivation on healthy lifestyle and glycemic control in diabetes patients. Participants will be randomized to two groups, the control group gets informational text message and the intervention group gets motivational SMS. The patients get a weekly text message and after 26 weeks the HbA1c and quality of life will be assessed.

DETAILED DESCRIPTION:
The investigators will examine the influence of increasing motivation on healthy lifestyle and glycemic control in diabetes patients. Participants will provide demographic and clinical information, fill human value questionnaires and quality of life questionnaires and decide on personal lifestyle-improvement goals. They will then be randomized to one of two groups: the control group gets informational text message and the intervention group gets motivational text message. The patients get a weekly text message and after 26 weeks we will check the HbA1c and quality of life. The text message will be personalized by including personal details acquired by a questionnaire. They will provide demographic and clinical information.

In addition, the influence of demographic characters and related DM character on the benefit of the motivational SMS will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled DM 2 patients (HbA1c > 8%)
* Know to read (Hebrew or Arabic)
* Have a cellular phone
* Can sign informed consent.

Exclusion Criteria:

* A life expectancy of less than one year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c levels at 6 months from beginning of messages | at 6 months from beginning of study
  Blood HbA1c levels are reflective of how well diabetes is controlled

SECONDARY OUTCOMES:
Diabetes Quality of Life questionnaire | at 6 months from beginning of study
  To design and test the reliability and validity of a brief treatment

CONTACTS AND LOCATIONS:
Overall Officials: Irit Hochberg, MD/PhD, Principal Investigator — Rambam Healthcare Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Text message program improves outcomes, decreases ED utilization among ED patients with poorly controlled diabetes. ED Manag. 2014 Feb;26(2):20-3. PMID 24505864
- [Background] Reinhardt JA, van der Ploeg HP, Grzegrzulka R, Timperley JG. lmplementing lifestyle change through phone-based motivational interviewing in rural-based women with previous gestational diabetes mellitus. Health Promot J Austr. 2012 Apr;23(1):5-9. doi: 10.1071/he12005. PMID 22730940
- [Background] Arora S, Peters AL, Agy C, Menchine M. A mobile health intervention for inner city patients with poorly controlled diabetes: proof-of-concept of the TExT-MED program. Diabetes Technol Ther. 2012 Jun;14(6):492-6. doi: 10.1089/dia.2011.0252. Epub 2012 Apr 23. PMID 22524591
- [Background] Hochberg I, Feraru G, Kozdoba M, Mannor S, Tennenholtz M, Yom-Tov E. Encouraging Physical Activity in Patients With Diabetes Through Automatic Personalized Feedback via Reinforcement Learning Improves Glycemic Control. Diabetes Care. 2016 Apr;39(4):e59-60. doi: 10.2337/dc15-2340. Epub 2016 Jan 28. No abstract available. PMID 26822328
- [Background] Ramachandran A, Snehalatha C, Ram J, Selvam S, Simon M, Nanditha A, Shetty AS, Godsland IF, Chaturvedi N, Majeed A, Oliver N, Toumazou C, Alberti KG, Johnston DG. Effectiveness of mobile phone messaging in prevention of type 2 diabetes by lifestyle modification in men in India: a prospective, parallel-group, randomised controlled trial. Lancet Diabetes Endocrinol. 2013 Nov;1(3):191-8. doi: 10.1016/S2213-8587(13)70067-6. Epub 2013 Sep 11. PMID 24622367